CLINICAL TRIAL: NCT01196299
Title: Prognostic Value of MR Imaging Markers in the Assessment of Traumatic Brain Injury Patients
Brief Title: Imaging of Traumatic Brain Injury
Acronym: Imaging of TBI
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Rao P Gullapalli, Professor, University of Maryland, Baltimore
Other Study IDs: HP-00040713; W81XWH-08-1-0725 (Other Grant/Funding Number: USA Med Research and Materiel Command)
Record Dates: First submitted 2010-09-03; First posted 2010-09-08 (Estimated); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Traumatic Brain Injury
Keywords: diffusion tensor imaging; magnetic resonance spectroscopy; traumatic brain injury; Metabolite changes; Cerebral perfusion; Hemorrhagic burden
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Severe Traumatic Brain Injury Group: The severe traumatic brain injury group are patients admitted to the study with an admission GCS between 3 and 8.
- Moderate Head Injury Group: The moderate head injury group are patients admitted to the study with an admission GCS from 9 to 12.
- Mild Head Injury Group: The mild head injury group are patients admitted to the study with an admission GCS from 13 to 15.
- Healthy Volunteer Group: Healthy volunteers will be selected to match the age distribution of the TBI groups. They must be absent of any abnormal radiological findings.

SUMMARY:
This project aims to study the prognostic ability of various MRI imaging markers in the evaluation of TBI patients. Cognitive, social, and occupational recovery will be measured at each time point, and compared to MRI findings. Healthy volunteers will serve as a comparison to the TBI patients.

It is hypothesized that novel MRI markers of metabolism, hemodynamics, functional connectivity, and tissue microstructure will be related to the clinical status of the patient, as well as their social and occupational outcomes.

DETAILED DESCRIPTION:
The goal of this study is to identify advanced magnetic resonance imaging markers that can serve as a prognostic marker in the evaluation and management of traumatic brain injury patients.

Magnetic resonance imaging and cognitive testing (when possible) will be performed in the acute (within 10 days following injury), and recovery stages (about 1 month, about 6 months,and about 18 months). The relationship between the advanced magnetic resonance imaging markers and the clinical condition of the patient will be evaluated at each time point to determine which combination of imaging markers best describe the current clinical status of the patient and which markers best predict a patient's outcome status.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Evidence of external head injury or facial trauma, or mechanism of injury consistent with brain trauma, including loss of consciousness or altered mental status.
* Residence within 90 minutes driving time of University of Maryland Medical Center, and willingness to attend follow-up appointments.

Exclusion Criteria:

* History of white matter disease or neurodegenerative disorders including Multiple Sclerosis, Huntington's Disease, Alzheimer's Disease, or Pick's Disease.
* History of Stroke
* History of treatment or diagnosis of psychiatric conditions: Major Depressive Disorder (MDD), Bipolar Disorder (BPD), Schizophrenia, or Dementia of any type.
* History of Brain Tumor
* Status post trauma due to asphyxiation
* Preexisting contraindications for Magnetic Resonance Imaging (MRI)
* Active Duty Military Status
* Police custody or prisoner status
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted with head trauma ranging from mild to severe.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2010-03-21 (Actual); Primary Completion 2015-04-17 (Actual); Study Completion 2015-09-05 (Actual)

PRIMARY OUTCOMES:
Identification of advanced MR imaging markers | 18 months post-injury
  Systematically study the imaging markers obtained from novel MRI techniques (diffusion tensor imaging (DTI), susceptibility-weighted imaging (SWI), MR spectroscopy, resting state MRI, and arterial spin labeling) and assess the markers for sensitivity.

SECONDARY OUTCOMES:
level of cognitive function | 18 months post-injury
extent of disability | 18 months post-injury
level of orientation | 18 months post-injury
level of functional independence | 18 months post-injury

CONTACTS AND LOCATIONS:
Overall Officials: Rao P Gullapalli, PhD, Principal Investigator — University of Maryland Medical School
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States